CLINICAL TRIAL: NCT04757610
Title: A Phase 3, Multicentre, Double-masked, Randomised Study to Evaluate the Efficacy and Safety of Intravitreal OPT-302 in Combination With Ranibizumab, Compared With Ranibizumab Alone, in Participants With nAMD
Brief Title: OPT-302 With Ranibizumab in Neovascular Age-related Macular Degeneration (nAMD)
Acronym: ShORe
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The primary endpoint was not achieved in the study.
Sponsor: Opthea Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPT-302-1004
Record Dates: First submitted 2021-02-12; First posted 2021-02-17 (Actual); Results first posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-06

CONDITIONS: Neovascular Age-related Macular Degeneration
MeSH Terms: interventions — Ranibizumab; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 0.5 mg ranibizumab with Standard Dosing 2.0 mg OPT-302 (Experimental): 0.5 mg ranibizumab intravitreal injection administered at 4-weekly intervals.
  2.0 mg OPT-302 intravitreal injection administered at 4-weekly intervals.
  Interventions: Biological: 2.0 mg OPT-302; Biological: 0.5 mg ranibizumab
- 0.5 mg ranibizumab with Extended Dosing 2.0 mg OPT-302 (Experimental): 0.5 mg ranibizumab intravitreal injection administered at 4-weekly intervals.
  2.0 mg OPT-302 intravitreal injection administered at 4-weekly intervals for three treatments, and then at 8-weekly intervals, with sham intravitreal injection administered at visits when OPT-302 is not.
  Interventions: Biological: 2.0 mg OPT-302; Biological: 0.5 mg ranibizumab
- 0.5 mg ranibizumab with sham (Sham Comparator): 0.5 mg ranibizumab intravitreal injection administered at 4-weekly intervals.
  Sham intravitreal injection administered at 4-weekly intervals.
  Interventions: Biological: 0.5 mg ranibizumab; Procedure: Sham

INTERVENTIONS:
Biological: 2.0 mg OPT-302 — intravitreal injection
  Arms: 0.5 mg ranibizumab with Extended Dosing 2.0 mg OPT-302; 0.5 mg ranibizumab with Standard Dosing 2.0 mg OPT-302
Biological: 0.5 mg ranibizumab — intravitreal injection
Procedure: Sham — intravitreal injection
  Arms: 0.5 mg ranibizumab with sham

SUMMARY:
A 2-year, phase 3, multicentre, randomised, parallel-group, sham-controlled, double-masked study. Primary efficacy will be determined at Week 52.

ELIGIBILITY:
Inclusion Criteria:

* Active subfoveal CNV lesion or juxtafoveal CNV lesion with foveal involvement that is secondary to AMD in the Study Eye.
* An ETDRS BCVA score between 60 and 25 (inclusive) letters in the Study Eye.

Main Exclusion Criteria:

* Any previous treatment for neovascular AMD.
* Clinically significant ocular disorders (other than neovascular AMD), which may interfere with assessment of BCVA, assessment of safety, or fundus imaging.
* Any current (or history of a) social, psychological, or medical condition that precludes enrolment into the study.

  * additional inclusion/exclusion criteria may apply

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 986 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (171):
- United States (70):
  - ShORe Investigational Site, Phoenix, Arizona
  - ShORe Investigational Site, Tucson, Arizona
  - ShORe Investigational Site, Bakersfield, California
  - ShORe Investigational Site, Campbell, California
  - ShORe Investigational Site, Encino, California
  - ShORe Investigational Site, Fullerton, California
  - ShORe Investigational Site, Glendale, California
  - ShORe Investigational Site, Huntington Beach, California
  - ShORe Investigational Site, Laguna Hills, California
  - ShORe Investigational Site, Long Beach, California
  - ShORe Investigational Site, Los Angeles, California
  - ShORe Investigational Site, Mountain View, California
  - ShORe Investigational Site, Palm Desert, California
  - ShORe Investigational site, Pasadena, California
  - ShORe Investiagtional Site, Poway, California
  - ShORe Investigational Site, Redlands, California
  - ShORe Investigational Site, Sacramento, California
  - ShORe Investigational Site, Santa Ana, California
  - ShORe Investigational Site, Torrance, California
  - ShORe Investigational Site, Colorado Springs, Colorado
  - ShORe Investigational Site, Denver, Colorado
  - ShORe Investigational Site, Lakewood, Colorado
  - ShORe Investigational Site, Longmont, Colorado
  - ShORe Investigational Site, Clearwater, Florida
  - ShORe Investigational Site, Fort Lauderdale, Florida
  - ShORe Investigational Site, Fort Myers, Florida
  - ShORe Investigational Site, Gainesville, Florida
  - ShORe Investigational Site, Lakeland, Florida
  - ShORe Investigational Site, Pensacola, Florida
  - ShORe Investigational Site, Pinellas Park, Florida
  - ShORe Investigational Site, Temple Terrace, Florida
  - ShORe Investigational Site, Augusta, Georgia
  - ShORe Investigational Site, Sandy Springs, Georgia
  - ShORe Investigational Site, Lemont, Illinois
  - ShORe Investigational Site, Indianapolis, Indiana
  - ShORe Investigational Site, Baltimore, Maryland
  - ShORe Investigational Site, Hagerstown, Maryland
  - ShORe Investigational Site, Towson, Maryland
  - ShORe Investigational Site, Springfield, Massachusetts
  - ShORe Investigational Site, Minneapolis, Minnesota
  - ShORe Investigational Site, St Louis, Missouri
  - ShORe Investigational Site, Reno, Nevada
  - ShORe Investigational Site, Bloomfield, New Jersey
  - ShORe Investigational Site, Toms River, New Jersey
  - ShORe Investigational Site, Hauppauge, New York
  - ShORe Investigational Site, Liverpool, New York
  - ShORe Investigational Site, Wake Forest, North Carolina
  - ShORe Investigational Site, Fargo, North Dakota
  - ShORe Investigational Site, Edmond, Oklahoma
  - ShORe Investigational Site, Tulsa, Oklahoma
  - ShORe Investigational Site, Eugene, Oregon
  - ShORe Investigational Site, Portland, Oregon
  - ShORe Investigational Site, Salem, Oregon
  - ShORe Investigational Site, Erie, Pennsylvania
  - ShORe Investigational Site, Beaufort, South Carolina
  - ShORe Investigational Site, Ladson, South Carolina
  - ShORe Investigational Site, Nashville, Tennessee
  - ShORe Investigational Site, Arlington, Texas
  - ShORe Investigational Site, Austin, Texas
  - ShORe Investigational Site, Bellaire, Texas
  - ShORe Investigational Site, Dallas, Texas
  - ShORe Investigational Site, Houston, Texas
  - ShORe Investigational Site, Katy, Texas
  - ShORe Investigational Site, McAllen, Texas
  - ShORe Investigational Site, San Antonio, Texas
  - ShORe Investigational Site, Tyler, Texas
  - ShORe Investigational Site, Willow Park, Texas
  - ShORe Investigational Site, Salt Lake City, Utah
  - ShORe Investigational Site, Charlottesville, Virginia
  - ShORe Investigational Site, Lynchburg, Virginia
- Argentina (6):
  - ShORe Investigational Site, Capital Federal, Ciudad Autonoma Buenos Aires
  - ShORe Investigational Site, Rosario, Santa Fe Province
  - ShORe Investigational Site, Rosario, Sante Fe
  - ShORe Investigational Site, Buenos Aires
  - ShORe Investigational Site, Ciudad Autonoma de Buenos Aire
  - ShORe Investigational Site, Córdoba
- Australia (2):
  - ShORe Investigational Site, Hurstville, New South Wales
  - ShORe Investigational Site, Melbourne, Victoria
- Brazil (6):
  - ShORe Investigational Site, Vitória, Cordoba
  - ShORe Investigational Site, Goiânia, Goiás
  - ShORe Investigational Site, Faxinal do Soturno, Rio Grande do Sul
  - ShORe Investigational site, Blumenau, Santa Catarina
  - ShORe Investigational Site, Santo André, São Paulo
  - ShORe Investigational Site, São Paulo
- ShORe Investigational Site, Sofia, Bulgaria
- Canada (3):
  - ShORe Investigational Site, Calgary, Alberta
  - ShORe Investigational Site, Edmonton, Alberta
  - ShORe Investigational Site, Mississauga, Ontario
- ShORe Investigational Site, Medellín, Colombia
- Czechia (3):
  - ShORe Investigational Site, Pardubice
  - ShORe Investigational Site, Prague
  - ShORe Investigational Site, Sokolov
- Denmark (3):
  - ShORe Investigational Site, Aarhus
  - ShORe Investigational Site, Glostrup Municipality
  - ShORe Investigational Site, Sønderborg
- France (4):
  - ShORe Investigational Site, Nice, Alpes-Maritimes
  - ShORe Investigational Site, Strasbourg, Bas Rhin
  - ShORe Investigational Site, Écully, Rhone
  - ShORe Investigational Site, Créteil, Val de Marr
- Germany (8):
  - ShORe Investigational Site, Ulm, Baden Wuerttermberg
  - ShORe Investigational Site, Heidelberg, Baden-Wurttemberg
  - ShORe Investigational Site, Goettigen, Lower Saxony
  - ShORe Investigational Site, Düsseldorf, Nordrhein
  - ShORe Investigational Site, Münster, Nordrhein
  - ShORe Investigational Site, Bonn, North Rhine-Westphalia
  - ShORe Investigational Site, Münster, North Rhine-Westphalia
  - ShORe Investigational Site, Hamburg
- Greece (3):
  - ShORe Investigational Site, Athens
  - ShORe Investigational Site, Ioannina
  - ShORe Investigational Site, Pátrai
- Hungary (3):
  - ShORe Investigational Site, Budapest
  - ShORe Investigational Site, Miskolc
  - ShORe Investigational Site, Szombathely
- India (9):
  - ShORe Investigational Site, Ahmedabad, Gujarat
  - ShORe Investigational Site, Surat, Gujarat
  - ShORe Investigational Site, Bangalore, Karnataka
  - ShORe Investigational Site, Pune, Maharashtra
  - ShORe Investigational Site, Chandigarh, Punjab
  - ShORe Investigational Site, Coimbatore, Tamil Nadu
  - ShORe Investigational Site, Lucknow, Uttar Pradesh
  - ShORe Investigational Site, Kolkata, West Bengal
  - ShORe Investigational Site, Mysuru
- Israel (5):
  - ShORe Investigational Site, Beersheba
  - ShORe Investigational Site, Haifa
  - ShORe Investigational Site, Kfar Saba
  - ShORe Investigational Site, Petah Tikva
  - ShORe Investigational Site, Rishon LeZiyyon
- Italy (7):
  - ShORe Investigational Site, Catanzaro, Reggio Calabria
  - ShORe Investigational Site, Bologna
  - ShORe Investigational Site, Chieti
  - ShORe Investiagational Site, Genova
  - ShORe Investigational Site, Roma
  - ShORe Investigational Site, Siena
  - ShORe Investigational Site, Udine
- ShORe Investigational Site, Riga, Latvia
- Malaysia (3):
  - ShORe Investigational Site, Batu Caves, Selangor
  - ShORe Investigational Site, Shah Alam, Selangor
  - ShORe Investigational Site, Kuala Lumpur
- Poland (7):
  - ShORe Investigational Site, Gdansk
  - ShORe Investigational Site, Krakow
  - ShORe Investigational Site, Olsztyn
  - ShORe Investigational Site, Szczecin
  - ShORe Investigational Site, Tarnowskie Góry
  - ShORe Investigational Site, Warsaw
  - ShORe Investigational Site, Wroclaw
- South Korea (5):
  - ShORe Investigational Site, Seongnam-si, Gyeonggi-do
  - ShORe Investigational Site, Daegu, Gyeongsangbuk-do
  - ShORe Investigational Site, Busan
  - ShORe Investigational Site, Gwangju
  - ShORe Investigational Site, Seoul
- Spain (9):
  - ShORe Investigational Site, Sant Cugat del Vallès, Barcelona
  - ShORe Investigational Site, Alcalá de Henares, Madrid
  - ShORe Investigational Site, Pamplona, Navarre
  - ShORe Investigational Site, Burjassot, Valencia
  - ShORe Investigational Site, Barcelona
  - ShORe Investigational Site, Burgos
  - ShORe Investigational Site, Córdoba
  - ShORe Investigational Site, Madrid
  - ShORe Investigational Site, Valencia
- Thailand (4):
  - ShORe Investigational Site, Pathum Wan, Bangkok
  - ShORe Investigational Site, Chiang Mai
  - ShORe Investigational Site, Khon Kaen
  - ShORe Investigational Site, Pathum Thani
- ShORe Investigational Site, Kiev, Ukraine
- United Kingdom (7):
  - ShORe Investigational Site, Crewe, Cheshire
  - ShORe Investigational Site, Southampton, Hampshire
  - ShORe Investigational Site, Leicester, Leicestershire
  - ShORe Investigational Site, Bristol, Somerset
  - ShORe Investigational Site, Guildford, Surrey
  - ShORe Investigational Site, Wolverhampton, West Midlands
  - ShORe Investigational Site, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants 50 years or older with active subfoveal CNV lesion or juxtafoveal CNV lesion with foveal involvement that is secondary to AMD in the study eye with an ETDRS BCVA score between 60 and 25 (inclusive) letters in the study eye.
Pre-assignment Details: Participants who met all inclusion criteria and none of the exclusion criteria were enrolled in the study.
  1 subject (in the 0.5 mg ranibizumab with standard dosing 2.0 mg OPT-302 arm) was enrolled, but never treated.
Groups:
- 0.5 mg Ranibizumab With Standard Dosing 2.0 mg OPT-302: 0.5 mg ranibizumab intravitreal injection (0.05mL) followed by 2.0 mg OPT-302 intravitreal injection (0.05mL) administered into the study eye at 4-weekly intervals through Week 96.
  2.0 mg OPT-302: intravitreal injection
  0.5 mg ranibizumab: intravitreal injection
- 0.5 mg Ranibizumab With Extended Dosing 2.0 mg OPT-302: 0.5 mg ranibizumab intravitreal injection (0.05mL) followed by 2.0 mg OPT-302 intravitreal injection (0.05mL) administered into the study eye at 4-weekly intervals for three treatments, and then at 8-weekly intervals through Week 96, with ranibizumab intravitreal injection followed by sham intravitreal injection administered into the study eye at the alternating visits when OPT-302 was not administered.
  2.0 mg OPT-302: intravitreal injection
  0.5 mg ranibizumab: intravitreal injection
  Sham: intravitreal injection
- 0.5 mg Ranibizumab With Sham: 0.5 mg ranibizumab intravitreal injection (0.05mL) followed by sham intravitreal injection administered into the study eye at 4-weekly intervals through Week 96.
  0.5 mg ranibizumab: intravitreal injection
  Sham: intravitreal injection
Period: Overall Study
Arm/Group | 0.5 mg Ranibizumab With Standard Dosing 2.0 mg OPT-302 | 0.5 mg Ranibizumab With Extended Dosing 2.0 mg OPT-302 | 0.5 mg Ranibizumab With Sham
Started (The number of participants randomized into the study) | 329 | 326 | 331
Treated (The number of participants randomized and treated) | 328 | 326 | 331
Completed (The number of participants that completed Week 100) | 167 | 168 | 171
Not Completed | 162 | 158 | 160
Not completed — Adverse Event | 13 | 10 | 5
Not completed — Death | 5 | 13 | 8
Not completed — Lack of Efficacy | 1 | 2 | 3
Not completed — Lost to Follow-up | 7 | 2 | 7
Not completed — Physician Decision | 4 | 1 | 2
Not completed — Withdrawal by Subject | 26 | 25 | 25
Not completed — Study Terminated by Sponsor | 105 | 105 | 110
Not completed — Randomized in Error | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-Treat (mITT) dataset comprised all randomised participants with at least one dose of study medication. Participants were analysed according to the study medication to which they were randomised for all efficacy analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.5 mg Ranibizumab With Standard Dosing 2.0 mg OPT-302 | 0.5 mg Ranibizumab With Extended Dosing 2.0 mg OPT-302 | 0.5 mg Ranibizumab With Sham | Total
Number analyzed (Participants) | 328 | 326 | 331 | 985
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 31 | 38 | 35 | 104
  >=65 years | 297 | 288 | 296 | 881
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.3 (8.28) | 75.8 (8.62) | 75.1 (8.52) | 75.4 (8.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 184 | 169 | 179 | 532
  Male | 144 | 157 | 152 | 453
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity is only captured in the United States
  Participants
    Hispanic or Latino | 10 | 10 | 5 | 25
    Not Hispanic or Latino | 117 | 121 | 123 | 361
    Unknown or Not Reported | 201 | 195 | 203 | 599
Race (NIH/OMB) [Count of Participants; unit: Participants] — A participant can be considered in more than one race category
  Participants
    American Indian or Alaska Native | 0 | 0 | 1 | 1
    Asian | 44 | 42 | 48 | 134
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 2
    Black or African American | 1 | 0 | 1 | 2
    White | 277 | 273 | 274 | 824
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 6 | 10 | 6 | 22
Early Treatment Retinopathy Study (ETDRS) Best-Corrected Visual Acuity (BCVA) Letters [Mean (Standard Deviation); unit: letters read] — The Early Treatment Retinopathy Study (ETDRS) Best-Corrected Visual Acuity (BCVA) letter score at baseline in the study eye.
  letters read | 52.1 (9.45) | 52.1 (8.83) | 52.5 (9.13) | 52.23 (9.14)
Choroidal Neovascularisation (CNV) Area by Fluorescein Angiography (FA) [Mean (Standard Deviation); unit: mm^2] — The Choroidal Neovascularisation (CNV) Area by Fluorescein Angiography (FA) at baseline.
  mm^2 | 6.256 (2.8634) | 6.576 (3.2278) | 6.286 (3.1770) | 6.373 (3.0894)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Early Treatment Diabetic Retinopathy Study (ETDRS) Best-corrected Visual Acuity (BCVA) Letters
Description: To determine the efficacy of intravitreal 2.0 mg OPT-302 when administered in combination with intravitreal 0.5 mg ranibizumab, in participants with neovascular age-related macular degeneration (nAMD), in terms of change in ETDRS BCVA letter score in the study eye from Baseline to Week 52. The primary analysis presented used mixed model for repeated measures in the overall population. (A positive outcome measure means an improvement in ETDRS BCVA letter score from baseline; a negative outcome measure means a deterioration in ETDRS BCVA letter score from baseline)
Time Frame: Baseline to Week 52
Population: Modified Intent-to-Treat (mITT) analysis set - comprised all randomised participants with at least one dose of study medication. Participants were analysed according to the study medication to which they were randomised for all efficacy analyses.
Measure: Least Squares Mean (Standard Error); unit: Letters read
Arm/Group | 0.5 mg Ranibizumab With Standard Dosing 2.0 mg OPT-302 | 0.5 mg Ranibizumab With Extended Dosing 2.0 mg OPT-302 | 0.5 mg Ranibizumab With Sham
Number analyzed (Participants) | 328 | 326 | 331
Letters read | 13.20 (0.728) | 12.41 (0.731) | 14.30 (0.719)
Statistical Analysis 1: Comparison: 0.5 mg Ranibizumab With Standard Dosing 2.0 mg OPT-302 vs 0.5 mg Ranibizumab With Sham; Test type: Superiority; p = 0.284421, MMRM; Least Squares Mean Difference = -1.10, 95% CI 2-sided [-3.10 to 0.91], Standard Error of Mean 1.023
Statistical Analysis 2: Comparison: 0.5 mg Ranibizumab With Extended Dosing 2.0 mg OPT-302 vs 0.5 mg Ranibizumab With Sham; Test type: Superiority; p = 0.066678, MMRM; Least Squares Mean Difference = -1.88, 95% CI 2-sided [-3.90 to 0.13], Standard Error of Mean 1.025

2. Secondary Outcome: Participants Gaining 15 or More ETDRS BCVA Letters
Description: To determine the effects of intravitreal 2.0 mg OPT-302 when administered in combination with intravitreal 0.5 mg ranibizumab, in participants with neovascular age-related macular degeneration (nAMD), in terms of proportion of participants gaining 15 or more letters in ETDRS BCVA in the study eye from Baseline to Week 52.
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 0.5 mg Ranibizumab With Standard Dosing 2.0 mg OPT-302 | 0.5 mg Ranibizumab With Extended Dosing 2.0 mg OPT-302 | 0.5 mg Ranibizumab With Sham
Number analyzed (Participants) | 292 | 290 | 297
Participants | 159 | 135 | 164

3. Secondary Outcome: Participants Gaining 10 More ETDRS BCVA Letters
Description: To determine the effects of intravitreal 2.0 mg OPT-302 when administered in combination with intravitreal 0.5 mg ranibizumab, in participants with neovascular age-related macular degeneration (nAMD), in terms of proportion of participants gaining 10 or more letters in ETDRS BCVA in the study eye from Baseline to Week 52.
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 0.5 mg Ranibizumab With Standard Dosing 2.0 mg OPT-302 | 0.5 mg Ranibizumab With Extended Dosing 2.0 mg OPT-302 | 0.5 mg Ranibizumab With Sham
Number analyzed (Participants) | 292 | 290 | 297
Participants | 198 | 182 | 202

4. Secondary Outcome: Change in Choroidal Neovascularisation (CNV) Area by Fluorescein Angiography (FA)
Description: To determine the effects of intravitreal 2.0 mg OPT-302 when administered in combination with intravitreal 0.5 mg ranibizumab, in participants with neovascular age-related macular degeneration (nAMD), in terms of change in CNV area as measured by FA in the study eye from Baseline to Week 52.
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mm^2
Arm/Group | 0.5 mg Ranibizumab With Standard Dosing 2.0 mg OPT-302 | 0.5 mg Ranibizumab With Extended Dosing 2.0 mg OPT-302 | 0.5 mg Ranibizumab With Sham
Number analyzed (Participants) | 147 | 132 | 154
mm^2 | -3.359 (0.3483) | -3.901 (0.3972) | -3.238 (0.3588)

5. Secondary Outcome: Participants With Absence of Both Sub-retinal Fluid and Intra-retinal Cysts by SD-OCT
Description: To determine the effects of intravitreal 2.0 mg OPT-302 when administered in combination with intravitreal 0.5 mg ranibizumab, in participants with neovascular age-related macular degeneration (nAMD), in terms of proportion of participants with absence of both sub-retinal fluid and intra-retinal cysts by SD-OCT in the study eye at Week 52.
Time Frame: at Week 52
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 0.5 mg Ranibizumab With Standard Dosing 2.0 mg OPT-302 | 0.5 mg Ranibizumab With Extended Dosing 2.0 mg OPT-302 | 0.5 mg Ranibizumab With Sham
Number analyzed (Participants) | 260 | 258 | 265
Participants | 33 | 22 | 22

ADVERSE EVENTS:
Time Frame: From Baseline to Week 100
Description: The safety dataset comprised all participants in the mITT dataset (all randomised participants with at least one dose of study medication). Participants were analysed according to the study medication received for all safety analyses. For Other (Not Including Serious) Adverse Events (AEs), non-serious AEs with a frequency greater than 5% within at least one arm are reported; the Total Affected is the total number of participants experiencing at least one non-serious TEAE during the study.
Arm/Group | 0.5 mg Ranibizumab With Standard Dosing 2.0 mg OPT-302 | 0.5 mg Ranibizumab With Extended Dosing 2.0 mg OPT-302 | 0.5 mg Ranibizumab With Sham
All-Cause Mortality (participants affected / at risk) | 5/328 | 13/327 | 8/330
Serious Adverse Events (participants affected / at risk) | 65/328 | 60/327 | 52/330
Other Adverse Events (participants affected / at risk) | 290/328 | 261/327 | 265/330
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.5 mg Ranibizumab With Standard Dosing 2.0 mg OPT-302 (N=328) | 0.5 mg Ranibizumab With Extended Dosing 2.0 mg OPT-302 (N=327) | 0.5 mg Ranibizumab With Sham (N=330)
Cataract (Eye disorders) | 3 (3) | 0 (0) | 0 (0)
Angle closure glaucoma (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Rhegmatogenous retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Retinal artery embolism (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vitritis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal pigment epithelial tear (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Eye inflammation (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Optic neuropathy (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal tear (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Endophthalmitis (Infections and infestations) | 4 (4) | 1 (1) | 1 (1) — Includes 1 non-study eye event in the Standard Dosing arm
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — Non-study eye event
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 3 (3) | 2 (3) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 3 (4) | 1 (1)
Coronary artery disease (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 6 (7) | 2 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal compartment syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Enterocele (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatic mass (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mesenteric arterial occlusion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis obstructive (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 3 (3) | 2 (2)
COVID-19 (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
COVID-19 Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Klebsiella urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Medical device site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
Craniofacial fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Femure fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Carotid artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperammonaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Type I diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Marginal zone lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Colorectal cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cutaneous T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 2 (2) | 3 (3)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 1 (2) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral thrombosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nerve compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neurodegenerative disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Rapid eye movement sleep behaviour disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary amyloidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertensive urgency (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral venous disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Venous hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.5 mg Ranibizumab With Standard Dosing 2.0 mg OPT-302 (N=328) | 0.5 mg Ranibizumab With Extended Dosing 2.0 mg OPT-302 (N=327) | 0.5 mg Ranibizumab With Sham (N=330)
Cataract (Eye disorders) | 39 (42) | 33 (35) | 14 (14)
Conjunctival haemorrhage (Eye disorders) | 32 (49) | 42 (61) | 24 (39)
Eye pain (Eye disorders) | 32 (70) | 19 (38) | 20 (29)
Vitreous floaters (Eye disorders) | 23 (25) | 21 (22) | 14 (15)
Vitreous detachment (Eye disorders) | 20 (20) | 16 (16) | 13 (13)
Intraocular pressure increased (Investigations) | 35 (93) | 29 (71) | 16 (34)
Neovascular age-related macular degeneration (Eye disorders) | 22 (24) | 19 (20) | 27 (29) — All events reported are in the non-study eye
Nasopharyngitis (Infections and infestations) | 57 (79) | 42 (64) | 39 (53)
COVID-19 (Infections and infestations) | 32 (32) | 27 (28) | 38 (39)
Urinary tract infection (Infections and infestations) | 22 (25) | 23 (30) | 20 (27)
Influenza (Infections and infestations) | 19 (22) | 12 (13) | 11 (11)
Upper respiratory tract infection (Infections and infestations) | 19 (25) | 11 (16) | 14 (18)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (26) | 23 (37) | 16 (22)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (15) | 15 (18) | 21 (25)
Headache (Nervous system disorders) | 21 (44) | 22 (32) | 25 (38)
Hypertension (Vascular disorders) | 19 (20) | 21 (25) | 27 (31)

LIMITATIONS AND CAVEATS:
This study was terminated early by the Sponsor because the study did not meet the primary endpoint. Thus, not all participants in this study completed the full duration of treatment.

Due to clinical program termination, data reported were not held to the expected standards for data verification and cleaning and are reported to the best of the Sponsor's ability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The principles for publication of results of this study will be addressed in clinical trial agreements between Opthea (Sponsor) and the study site, and Opthea and the subcontractors performing the study. Results means any and all information and know-how (whether patentable or not) which is discovered, invented or developed or which arises in the course of or as a result of the conduct of the Study, including any and all improvements to the products being studied.

DOCUMENTS (2):
  • Study Protocol (2023-12-19): https://cdn.clinicaltrials.gov/large-docs/10/NCT04757610/Prot_001.pdf
  • Statistical Analysis Plan (2023-12-19): https://cdn.clinicaltrials.gov/large-docs/10/NCT04757610/SAP_002.pdf